CLINICAL TRIAL: NCT06587217
Title: Neurobiological Drivers of Mobility Resilience: The Dopaminergic System
Brief Title: Neurobiological Drivers of Mobility Resilience: The Dopaminergic System - Supplemental Open-Label Arm
Acronym: RES
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Principal Investigator, Chatkaew Pongmala, Research Investigator, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: HUM00156490-B; 5U01AG061393-05 (NIH)
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Parkinsonian Signs in Older Persons
Keywords: slow gait; Parkinsonian signs
MeSH Terms: interventions — Carbidopa; carbidopa, levodopa drug combination

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Carbidopa Monotherapy and Carbidopa-Levodopa (Experimental): Participants will begin by taking 25mg of Carbidopa monotherapy three times per day (TID) for 3 days. On day four, participants will begin taking 1 tablet of Carbidopa-Levodopa (25/100mg) TID in addition to the Carbidopa monotherapy. On day seven, participants will increase to 1.5 tablets of Carbidopa-Levodopa (25/100mg) TID while maintaining 25mg Carbidopa monotherapy TID. The intervention will end after ten days of supplementation.
  Interventions: Drug: Carbidopa 25 mg; Drug: Carbidopa-Levodopa 25/100 mg

INTERVENTIONS:
Drug: Carbidopa 25 mg — Participants will take one 25mg Carbidopa tablet 3 times a day for 10 days.
Drug: Carbidopa-Levodopa 25/100 mg — Participants will take one 25/100mg carbidopa-levodopa tablet 3 times a day on days 4-6, then increase to 1.5 tablets 3 times a day on days 7-10.
  Other Names: Sinemet

SUMMARY:
Walking with age becomes both slower and less 'automated', requiring more attention and brain resources. As a result, older adults have a greater risk of negative outcomes and falls. There is an urgent need to identify factors that can help compensate for these harmful factors and reduce walking impairments, as there are currently no effective treatments available. Investigators have recently discovered that ~20% of older adults maintain fast walking speed even in the presence of small blood vessel brain changes and leg problems, thus appearing to be protected against these harmful factors. The investigators work suggests that the brain dopamine (DA) system may be a source of this protective capacity. Investigators have also shown that lower levels of dopamine are associated with slow walking. Investigators will be investigating the role of dopamine on slow walking and other parkinsonian signs in this open-label study using detailed clinical assessment, assessment of dopamine activity, and clinical interventions.

DETAILED DESCRIPTION:
Walking with age becomes both slower and less 'automated', requiring more attention and prefrontal resources. As a result, older adults have a greater risk of adverse mobility outcomes and falls. Walking disturbances in the elderly have been linked to changes in both cerebral, in particular small vessel disease (cSVD), and peripheral systems. There is an urgent need to identify factors that can help compensate for these harmful factors and reduce walking impairments, as there are currently no effective treatments available. Although effective mobility is the end result of the functional capacity of both central and peripheral systems, the brain's unique modulatory and adaptive capacity may provide clues for novel interventions. For example, investigators have recently discovered that ~20% of older adults maintain fast walking speed even in the presence of age related cSVD and peripheral system impairments, thus appearing resilient to these harmful factors. The investigators work suggests that the nigrostriatal dopamine (DA) system may be a source of this resilience. As investigators recent findings suggest, DA neurotransmission positively predicts walking speed; it also attenuates the negative effects of age related cSVD and peripheral system impairments on walking speed. These findings are consistent with post-mortem evidence that a combination of loss of nigral DA neurons and cSVD best predict age-related walking impairment. The nigrostriatal DA system plays a critical role in motor control; nigrostriatal. DA neurotransmission regulates the automated execution of overlearned motor tasks via its connections with sensorimotor cortical and subcortical areas.

The investigators hypothesize that higher nigrostriatal DA neurotransmission drives resilience to cSVD and peripheral system impairments, via higher connectivity of sensorimotor networks, thus increasing automaticity of walking and reducing prefrontal engagement while walking. Unlike cSVD and brain structural impairments, DA neurotransmission is potentially modifiable, thereby offering novel approaches to treat non-resilient elderly in a targeted fashion. This study is an arm of a previously completed translational pilot biomechanistic target engagement study in older adults with slow walking and/or parkinsonian signs (NCT04325503). This sub-study will further expand upon biomechanistic target engagement findings by increasing the sample size using an additional, open-label experimental design.

The study will include elderly men and women age 60 or older with evidence of mild parkinsonian signs (MPS, or slow gait (< 1m/s)).

ELIGIBILITY:
Inclusion Criteria:

* Age 60 or older (M/F)
* Evidence of mild parkinsonian signs (incl. slow gait (<1m/s))

Exclusion Criteria:

* Evidence of prior established diagnosis and/or treatment for PD.
* Presence of clinically significant degenerative joint disease and/or neuropathy interfering with proper assessment of the motor exam.
* Presence of significant dementia.
* History of stroke with residual clinical deficit interfering with walking.
* For optional MR imaging only: Participants in whom magnetic resonance imaging (MRI) is contraindicated including, but not limited to, those with a pacemaker, presence of metallic fragments near the eyes or spinal cord, or cochlear implant.
* For optional brain imaging only: Severe claustrophobia precluding neuroimaging procedures.
* Participants that have been on monoamine oxidase inhibitors (MAOIs) within 2 weeks prior to starting study.
* Inability to stand or walk without an assistive device
* Hypersensitivity to the carbidopa, levodopa, and tablet components.
* History of myocardial infarction (MI) with residual arterial, nodal or ventricular arrhythmia
* History of peptic ulcer
* Chronic wide angle glaucoma
* Narrow angle glaucoma
* Major psychotic disorder
* Severe cardiovascular or pulmonary disease, bronchial asthma, renal, hepatic or endocrine disease
* Subjects on dopamine D2 receptor antagonists, dopamine depleting agents, and metoclopramide.
* Any other medical history determined by investigators to preclude safe participation.

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2024-10-29 (Actual); Primary Completion 2025-04-03 (Actual); Study Completion 2025-04-03 (Actual)

PRIMARY OUTCOMES:
Average Gait Speed | Pre and Post 7-13 day intervention
  Average gait speed as measured using wearable sensors and while walking on a sensor mat. Measured in meters per second.

CONTACTS AND LOCATIONS:
Overall Officials: Chatkaew Pongmala, PhD, Principal Investigator — University of Michigan
Locations (2):
- United States (2):
  - Domino's Farms, Ann Arbor, Michigan
  - University Hospital, Ann Arbor, Michigan

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-12-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT06587217/Prot_SAP_000.pdf
  • Informed Consent Form (2025-04-17): https://cdn.clinicaltrials.gov/large-docs/17/NCT06587217/ICF_001.pdf